CLINICAL TRIAL: NCT01898091
Title: Randomized Controlled Double-blinded Clinical Trial of an Herbal Mouthrinse for Radiotherapy Induced Mucositis in Cancer Patients
Brief Title: Herbal Mouthrinse for Oral Mucositis Study
Acronym: OM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Susan G. Reed, Associate Professor, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 101529; 1R21CA158530-01A1 (NIH)
Record Dates: First submitted 2013-07-02; First posted 2013-07-12 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Oral Mucositis
Keywords: Oral; Mucositis; Stomatitis; Radiotherapy
MeSH Terms: conditions — Stomatitis; Mucositis | interventions — anise oil; Ascorbic Acid; Phosphatidylinositol 3-Kinases; Glycerol; peppermint oil; Poloxamer; Sorbic Acid; Water; Xylitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neem Mouthrinse (Experimental): Participants will rinse for 30 seconds with the measured 10ml dose of the assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Interventions: Drug: Neem Mouthrinse; Drug: Placebo Mouthrinse
- Placebo Mouthrinse (Placebo Comparator): Participants will rinse for 30 seconds with the measured 10ml dose of the assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Interventions: Drug: Placebo Mouthrinse

INTERVENTIONS:
Drug: Neem Mouthrinse — 10ml dose of assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Other Names: aloe; anise; ascorbic acid; clove; glycerin; extract of neem leaf; peppermint; poloxamer 407; potassium sorbate; spearmint; thyme; water; xylitol
  Arms: Neem Mouthrinse
Drug: Placebo Mouthrinse — 10ml dose of assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Other Names: aloe; anise; ascorbic acid; clove; glycerin; peppermint; poloxamer 407; potassium sorbate; spearmint; thyme; water; xylitol

SUMMARY:
This study involves adults receiving radiation therapy for head and neck cancer and will test whether or not the study mouthrinse may lessen oral mucositis.

DETAILED DESCRIPTION:
The broad goal of our research is development of an effective Complementary and Alternative Medicine (CAM) approach to prevent mucositis or lessen its severity and complications. Oral mucositis (OM) is a clinically challenging and debilitating side effect of conventional radiotherapy (RT), affecting almost all patients undergoing RT for head and neck cancer. OM includes inflammation of the oral mucosa with or without opportunistic microbial infection. It ranges from mild erythema to severe ulceration accompanied by persistent pain leading to inability to tolerate or swallow food and fluids. OM frequently causes unwanted cancer treatment dose reductions or breaks in therapy. Despite use of pain medications, severe OM is associated with substantially increased use of costly health care resources. Presently, there are no effective treatments for OM. The primary aim of the current proposal is to determine whether or not a mouthrinse containing an herbal extract with known anti-inflammatory and anti-microbial medicinal properties, will reduce the severity of oral mucositis in cancer patients undergoing conventional radiotherapy to the head and neck. Because of the prominent inflammatory and microbial aspects of OM we anticipate that the herbal mouthrinse will reduce the severity of the pain and secondary infections associated with OM, and will improve the quality of life in head and neck cancer patients undergoing RT. Therefore, the specific aims of our Phase II double-blind, randomized, controlled trial are 1) to determine if the severity of oral mucositis is reduced in RT patients receiving the herbal mouthrinse compared to patients receiving the comparison mouthrinse and 2) to determine the effects of the herbal mouthrinse on the microbial environment of the oral cavity and on quality of life. Findings from this study will provide evidence to support more in-depth biological assessment of the anti-inflammatory and anti-microbial mechanisms by which the herbal extract reduces oral mucositis, and additional study in other populations experiencing mucositis.

ELIGIBILITY:
Inclusion Criteria:

* Anatomic site: lip (inner aspect), oral cavity, pharynx or larynx; includes tonsils and salivary glands (ICD-9: 140-149 or 161).
* Malignant tumor: ICD-O morphology 2 (in situ) or 3 (malignant, invasive or infiltrating).
* Adult aged 18-89 years.
* Patient recommended or planned to undergo radiotherapy to the head and neck regions, as part of their cancer treatment regimen.
* Radiotherapy to be given in standard doses over a 4 - 7 week period.

Exclusion Criteria:

* Prior radiation treatment for cancer of the oral cavity, head or neck.
* Baseline mouth and throat soreness (MTS) extreme score of 4.
* Eastern Cooperative Oncology Group (ECOG) performance status >2.
* Unable to sign Informed Consent.
* Known history of allergy to any of the mouthrinse constituents (aloe, anise, ascorbic acid, clove, glycerin, peppermint, poloxamer 407, potassium sorbate, spearmint, thyme, water, xylitol).
* Inability to use a mouth rinse.
* Patient unable to communicate with study personnel in English (either themselves or an interpreter).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan G. Reed, DDS, DrPH, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After publication of the results of the primary and secondary endpoints of the trial, we will offer our collected experience to other interested clinicians/scientists. Our first priority is that any data sets that are used be subject of a confidentiality agreement. Any clinical data that is shared will be stripped of any subject personal information (de-indentified data). Our intent, if the trial results are promising is to share the findings through the HCC Clinical Trial Network. If our intervention is useful we are open to further investigation though clinical trial and other cooperative groups. Dr. Susan Reed, as PI, will participate in all sharing activities.

REFERENCES:
- [Result] Elting LS, Keefe DM, Sonis ST, Garden AS, Spijkervet FK, Barasch A, Tishler RB, Canty TP, Kudrimoti MK, Vera-Llonch M; Burden of Illness Head and Neck Writing Committee. Patient-reported measurements of oral mucositis in head and neck cancer patients treated with radiotherapy with or without chemotherapy: demonstration of increased frequency, severity, resistance to palliation, and impact on quality of life. Cancer. 2008 Nov 15;113(10):2704-13. doi: 10.1002/cncr.23898. PMID 18973181

RESULTS

PARTICIPANT FLOW:
Groups:
- Neem Mouthrinse: Participants will rinse for 30 seconds with the measured 10ml dose of the assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Neem Mouthrinse: 10ml dose of assigned study mouthrinse [mouthrinse base plus 1% solution by weight of neem supercritical extract], three times per day, for approximately 7 weeks during radiation therapy.
- Placebo Mouthrinse: Participants will rinse for 30 seconds with the measured 10ml dose of the assigned study mouthrinse, three times per day, for approximately 7 weeks during radiation therapy.
  Placebo Mouthrinse: 10ml dose of assigned study mouthrinse [mouthrinse base], three times per day, for approximately 7 weeks during radiation therapy.
Period: Overall Study
Arm/Group | Neem Mouthrinse | Placebo Mouthrinse
Started | 25 (Allocated to intervention. All allocated received intervention.) | 25 (Allocated to intervention. All allocated received intervention.)
Completed | 23 | 19
Not Completed | 2 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neem Mouthrinse | Placebo Mouthrinse | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.4) | 61 (11.5) | 59 (11.5)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 23 | 19 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 16 | 17 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 19 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Change in Mean Mouth and Throat Soreness (MTS) Score From Baseline Through Weeks of Radiation Therapy Using the MTS Question of the Modified Oral Mucositis Daily Questionnaire*.
Description: Severity is assessed as the maximum change in mean mouth and throat soreness (MTS) score from baseline during the weeks of RT, using MTS question of the validated Oral Mucositis Daily Questionnaire (modified OMDQ): "During the past 24 hours, how much mouth and throat soreness did you have?" The MTS score is a 5-point score, ranging from 0=No soreness to 4=Extreme soreness. We compared the maximum change in MTS score between the two groups using the Wilcoxon rank sum test with a one-sided alpha of 0.05.
Time Frame: MTS score is collected at the baseline visit and once each week during the 7 weeks of radiation therapy.
Population: Exclusion criterion was those with a baseline mouth and throat soreness (MTS) extreme score of 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Neem Mouthrinse | Placebo Mouthrinse
Number analyzed (Participants) | 23 | 19
units on a scale | 1.91 (1.34) | 1.47 (1.22)
Statistical Analysis 1: Comparison: Neem Mouthrinse vs Placebo Mouthrinse; Simulations determined power to detect significant difference defined as a mean difference of 1 unit (MTS scale). Feasibility study provided proportion of patients in control and neem group with change scores of 0, 1, 2, 3, and 4 as (5%, 10%, 10%, 45% and 30%) and (15%, 20%, 30%, 25% and 10%), respectively. Simulated 10,000 trials using multinomial distributions by the percentages above, with 20 patients per group, provided 80% power to detect 0.9 unit difference using a one-sided alpha of 0.05; Test type: Superiority or Other; p = 0.84, Wilcoxin rank sum test

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: All adverse events are reported. The population includes a total of 50 patients, which includes 8 patients who were not evaluable for major outcome results.
Arm/Group | Neem Mouthrinse | Placebo Mouthrinse
Serious Adverse Events (participants affected / at risk) | 1/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neem Mouthrinse (N=25) | Placebo Mouthrinse (N=25)
Respiratory insufficiency (General disorders) | 1 (1) | 0 (0) — Respiratory insufficiency; pneumonia, aspiration; shock, septic; stroke
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neem Mouthrinse (N=25) | Placebo Mouthrinse (N=25)
Exanthema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — External mouth transient rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No